CLINICAL TRIAL: NCT03793517
Title: Decitabine Plus mBU/CY for High Risk Acute Leukemia With Minimal Residual Disease Pre-HSCT
Brief Title: Decitabine Plus mBU/CY for High Risk Acute Leukemia With MRD Pre-HSCT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojun Huang,MD, Director of the Hematology Department, Peking University People's Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: decitabine pre-HSCT in MRD+ AL
Record Dates: First submitted 2018-12-23; First posted 2019-01-04 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Stem Cell Transplant Complications; Leukemia, Myeloid, Acute; Leukemia Relapse
Keywords: high risk acute myeloid leukemia; hematopoietic stem cell transplantation; leukemia relapse; preparation regimen; decitabine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Decitabine

STUDY DESIGN:
Intervention Model Description: Patients enrolled in this study would receive decitabine 200mg·m-2·d-1 on day -12 and -11 pre-HSCT. The conditioning therapy for human leukocyte antigen (HLA)-mismatched HSCT patients was modified BU/CY plus ATG. In matched sibling transplantations, patients received hydroxycarbamide (80 mg·kg-1) orally on day -10 and a lower dose of Ara-C (2 g·m-2·d-1) on day -9, but otherwise an identical regimen to the HLA-mismatched patients without ATG.BM samples from patients would be obtained to assess leukemia status after HSCT. The time points that we monitored BM samples included at time of allo-HSCT; 1 month, 2 months, 3 months, 4.5 months, 6 months, 9 months, and 12 months after allo-HSCT; and every 6 months thereafter to the defined endpoints or for at least until 5 year after transplantation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decitabine plus mBU/CY for HLA-mismatched HSCT (Experimental): Decitabine plus mBU/CY as precondition regimen for High Risk Acute Leukemia With MRD at the time of HLA-mismatched HSCT.
  Details:
  The conditioning therapy for human eukocyte antigen (HLA)-mismatched HSCT patients was decitabine plus modified BU/CY and ATG,consisting of decitabine 100mg·m-2·d-1 q12h on days-12 and -11,cytarabine (Ara-C 4 g·m-2·d-1) intravenously on days -10 to -9, busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, cyclophosphamide (CY 1.8 g·m-2·d-1), intravenously on days -5 to -4, simustine (Me-CCNU, 250 mg/m2), orally once on day -3, and ATG (2.5 mg·kg-1·d-1) intravenously on days -5 to -2.
  Interventions: Drug: Decitabine; Drug: mBU/CY and ATG
- Decitabine plus mBU/CY for matched sibling transplant (Experimental): Decitabine plus mBU/CY as precondition regimen for High Risk Acute Leukemia With MRD at the time of matched sibling transplant.
  Details:
  In matched sibling transplantations, patients received decitabine 100mg·m-2·d-1 q12h on days-12 and -11,hydroxycarbamide (80 mg/kg) orally on day -10 and a lower dose of Ara-C (2 g·m-2·d-1) on day -9, busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, cyclophosphamide (CY 1.8 g·m-2·d-1), intravenously on days -5 to -4, simustine (Me-CCNU, 250 mg/m2), orally once on day -3.
  Interventions: Drug: Decitabine; Drug: mBU/CY

INTERVENTIONS:
Drug: Decitabine — Decitabine 200mg.m-2.d-1 intervanously on days -12 and -11
Drug: mBU/CY and ATG — Ara-C 4 g·m-2·d-1 intravenously on days -10 to -9 Busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, Cyclophosphamide (CY 1.8 g·m-2·d-1) intravenously on days -5 to -4 Simustine (Me-CCNU, 250 mg·m-2) orally once on day -3 ATG (2.5 mg·kg-1·d-1) intravenously on days -5 to -2
  Arms: Decitabine plus mBU/CY for HLA-mismatched HSCT
Drug: mBU/CY — hydroxycarbamide (80 mg·kg-1) orally on day -10 Ara-C (2 g·m-2·d-1) on day -9 Busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, Cyclophosphamide (CY 1.8 g·m-2·d-1) intravenously on days -5 to -4 Simustine (Me-CCNU, 250 mg·m-2) orally once on day -3
  Arms: Decitabine plus mBU/CY for matched sibling transplant

SUMMARY:
Allogeneic haematopoietic stem cell transplantation (allo-HSCT) remains one of the currently available curative therapies for acute leukemia (AL). Leukemia relapse is one of the mainly causes of transplant failure. We reported previously that patients with high-risk molecular biomarkers who still have detectable minimal residual disease(MRD) pre-HSCT were at very high risk of relapse, with cumulative relapse rate of 50-80%. Decitabine has been demonstrated efficacy in the treatment of patients with recurrent or refractory leukemia and myelodysplastiv syndrome. It was reported that the combination of decitabine, with busufan and cyclophosphamide as a preparative regimen for allo-HSCT using HLA-matching donors was safe and effective. In this prospective, single-arm clinical trial, we aimed to examine the efficacy of combining decitabine with modified busulfan and cyclophosphamide (mBU/CY) as a preparative regimen for allo-HSCT in patients with very high-risk AL and detectable MRD pre-HSCT.

DETAILED DESCRIPTION:
Patients enrolled in this study would receive decitabine 200mg·m-2·d-1 on day -12 and -11 pre-HSCT. The conditioning therapy for human leukocyte antigen (HLA)-mismatched HSCT patients was modified BU/CY plus ATG (thymoglobulin; Sang Stat, France) consisting of cytarabine (Ara-C 4 g·m-2·d-1) intravenously on days -10 to -9, busulfan (BU 3.2 mg·kg-1·d-1) intravenously on days -8 to -6, cyclophosphamide (CY 1.8 g·m-2·d-1), intravenously on days -5 to -4, semustine (Me-CCNU, 250 mg·m-2), orally once on day -3, and ATG (2.5 mg·kg-1·d-1) intravenously on days -5 to -2. In matched sibling transplantations, patients received hydroxycarbamide (80 mg·kg-1) orally on day -10 and a lower dose of Ara-C (2 g·m-2·d-1) on day -9, but otherwise an identical regimen to the HLA-mismatched patients without ATG.

BM samples from patients were obtained to assess leukemia status after HSCT. The time points that we monitored BM samples included at time of allo-HSCT; 1 month, 2 months, 3 months, 4.5 months, 6 months, 9 months, and 12 months after allo-HSCT; and every 6 months thereafter to the defined endpoints or for at least until 5 years after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* acute leukemia patients with MLL-r,TLS-ERG,or SIL-TAL1,whose minimal residual disease were detectable pre-HSCT

Exclusion Criteria:

* pregnancy women
* uncontrolled severe infection

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
1 year cumulative incidence of relapse | 1 year post allo-HSCT
  The cumulative incidence of relapse at 1 year post allo-HSCT
2 year cumulative incidence of relapse | 2 years post allo-HSCT
  The cumulative incidence of relapse at 2 years post allo-HSCT

SECONDARY OUTCOMES:
Non-relapse mortality | 1 year post allo-HSCT
  The cumulative incidence of non-relapse mortality at 1 year post allo-HSCT
1 year overall survival | 1 year post allo-HSCT
  The overall survival at 1 year post allo-HSCT
5 years overall survival | 5 years post allo-HSCT
  The overall survival at 5 years post allo-HSCT
1 year leukemia free survival | 1 year post allo-HSCT
  The leukemia free survival at 1 years post allo-HSCT
5 years leukemia free survival | 5 years post allo-HSCT
  The leukemia free survival at 5 years post allo-HSCT
engraftment | 100 days post allo-HSCT
  The total neutrophil and platelet engraftment rate
Acute graft versus host disease | 100 days post allo-HSCT
  The cumulative incidence of grade II-IV acute graft versus host disease
Chronic graft versus host disease | 1 years post allo-HSCT
  The cumulative incidence of intermediate to severe chronic graft versus host disease

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jun Huang, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University Institute of Hematology,Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No